CLINICAL TRIAL: NCT03393377
Title: Preventive Arterial Wall Phenotype in Subjects at Moderate Cardiovascular Risk Induced by Very Low-dose Fluvastatin/Valsartan Combination: a Pilot Study
Brief Title: Preventive Arterial Wall Phenotype and Low-dose Fluvastatin/Valsartan Combination
Acronym: AGE-ZT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Martina Turk Veselič, Medical Doctor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGE-ZT
Record Dates: First submitted 2017-12-29; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Atherosclerosis
Keywords: arterial stiffness; endothelial dysfunction; fluvastatin; valsartan; inflammatory markers; oxidative stress; SIRT1
MeSH Terms: conditions — Atherosclerosis | interventions — Fluvastatin; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): received fluvastatin 10 mg and valsartan 20 mg (low-flu/val) for 30 days
  Interventions: Drug: fluvastatin 10 mg and valsartan 20 mg
- control group (Placebo Comparator): received placebo for 30 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluvastatin 10 mg and valsartan 20 mg
  Other Names: low-flu/val
  Arms: intervention group
Drug: placebo
  Arms: control group

SUMMARY:
The study was designed to test whether short-term treatment with a very low-dose combination of fluvastatin and valsartan could induce improvement of endothelial function, arterial stiffness, vascular inflammation, oxidative stress and expression of protective genes in subjects with moderate cardiovascular risk.

DETAILED DESCRIPTION:
The largest population that suffers from cardiovascular events are subjects at moderate cardiovascular risk. However, no effective and safe preventive treatment is available for this population. This study aimed to investigate whether their arterial wall phenotype could be turned to a preventive direction by low-dose fluvastatin/valsartan combination (low-flu/val).

Twenty males at moderate cardiovascular risk (as classified by SCORE) were blindly randomised into the intervention group (n=10, low-flu/val: 10 mg/20mg) or control group (n=10, placebo). At inclusion and after 30 days of treatment, brachial flow-mediated dilatation (FMD), beta stiffness coefficient, carotid pulse wave velocity (c-PWV), carotid-femoral PWV, reactive hyperaemia index, high-sensitivity C-reactive protein (hs-CRP), interleukin 6, vascular cell adhesion molecule 1, total antioxidant status and expression of several protective genes (SIRT1, mTOR, NF-κB1, NFE2L2, PRKAA1) were followed.

ELIGIBILITY:
Inclusion Criteria:

* moderate cardiovascular risk according to Systematic Coronary Risk Estimation (SCORE) risk charts of the European Society of Cardiology
* males
* aged between 40 and 55 years

Exclusion Criteria:

* diabetes mellitus
* manifest peripheral artery disease or carotid artery disease
* acute infection
* chronic diseases
* present therapy with fluvastatin and/or valsartan

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
brachial flow-mediated dilatation (FMD) | 30 days
  FMD measured by ultrasound on right brachial artery (as result of reactive hyperaemia)
reactive hyperaemia index (RHI) | 30 days
  RHI measured by Endopat device
beta stiffness coefficient | 30 days
  assessed by ultrasound employing e-Tracking on right common carotid artery
carotid pulse wave velocity (c-PWV) | 30 days
  assessed by ultrasound employing e-Tracking on right common carotid artery
carotid-femoral PWV (cf-PWV) | 30 days
  cf-PWV measured by Sphygmocor device
high-sensitivity C-reactive protein (hs-CRP) | 30 days
  inflammatory marker
interleukin 6 (IL-6) | 30 days
  inflammatory marker
vascular cell adhesion molecule 1 (VCAM1) | 30 days
  inflammatory marker
total antioxidant status (TAS) | 30 days
  marker of oxidative stress
gene SIRT1 | 30 days
  Hs01009006_m1
gene mTOR | 30 days
  Hs00234522_m1
gene NF-kB1 | 30 days
  Hs00765730_m1
gene Nrf2/NFE2L2 | 30 days
  Hs00975961_g1
gene AMPK/PRKAA1 | 30 days
  Hs01562315_m1

SECONDARY OUTCOMES:
brachial flow-mediated dilatation (FMD) | 10 weeks after treatment completion
  FMD measured by ultrasound on right brachial artery (as result of reactive hyperaemia)
reactive hyperaemia index (RHI) | 10 weeks after treatment completion
  RHI measured by Endopat device
beta stiffness coefficient | 10 weeks after treatment completion
  assessed by ultrasound employing e-Tracking on right common carotid artery
carotid pulse wave velocity (c-PWV) | 10 weeks after treatment completion
  assessed by ultrasound employing e-Tracking on right common carotid artery
carotid-femoral PWV (cf-PWV) | 10 weeks after treatment completion
  cf-PWV measured by Sphygmocor device

REFERENCES:
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Matsuzawa Y, Kwon TG, Lennon RJ, Lerman LO, Lerman A. Prognostic Value of Flow-Mediated Vasodilation in Brachial Artery and Fingertip Artery for Cardiovascular Events: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2015 Nov 13;4(11):e002270. doi: 10.1161/JAHA.115.002270. PMID 26567372
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Paneni F, Diaz Canestro C, Libby P, Luscher TF, Camici GG. The Aging Cardiovascular System: Understanding It at the Cellular and Clinical Levels. J Am Coll Cardiol. 2017 Apr 18;69(15):1952-1967. doi: 10.1016/j.jacc.2017.01.064. PMID 28408026
- [Background] Lunder M, Janic M, Jug B, Sabovic M. The effects of low-dose fluvastatin and valsartan combination on arterial function: a randomized clinical trial. Eur J Intern Med. 2012 Apr;23(3):261-6. doi: 10.1016/j.ejim.2011.11.011. Epub 2011 Dec 12. PMID 22385885
- [Background] Boncelj Svetek M, Erzen B, Kanc K, Sabovic M. Impaired endothelial function and arterial stiffness in patients with type 2 diabetes - The effect of a very low-dose combination of fluvastatin and valsartan. J Diabetes Complications. 2017 Mar;31(3):544-550. doi: 10.1016/j.jdiacomp.2016.12.002. Epub 2016 Dec 16. PMID 28012835
- [Background] Janic M, Lunder M, Prezelj M, Sabovic M. A combination of low-dose fluvastatin and valsartan decreases inflammation and oxidative stress in apparently healthy middle-aged males. J Cardiopulm Rehabil Prev. 2014 May-Jun;34(3):208-12. doi: 10.1097/HCR.0000000000000027. PMID 24263076
- [Background] Sosnowska B, Mazidi M, Penson P, Gluba-Brzozka A, Rysz J, Banach M. The sirtuin family members SIRT1, SIRT3 and SIRT6: Their role in vascular biology and atherogenesis. Atherosclerosis. 2017 Oct;265:275-282. doi: 10.1016/j.atherosclerosis.2017.08.027. Epub 2017 Aug 26. PMID 28870631
- [Background] Yusuf S, Bosch J, Dagenais G, Zhu J, Xavier D, Liu L, Pais P, Lopez-Jaramillo P, Leiter LA, Dans A, Avezum A, Piegas LS, Parkhomenko A, Keltai K, Keltai M, Sliwa K, Peters RJ, Held C, Chazova I, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Sanchez-Vallejo G, McKelvie R, Pogue J, Jung H, Gao P, Diaz R, Lonn E; HOPE-3 Investigators. Cholesterol Lowering in Intermediate-Risk Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2021-31. doi: 10.1056/NEJMoa1600176. Epub 2016 Apr 2. PMID 27040132
- [Background] Robinson JG, Gidding SS. Curing atherosclerosis should be the next major cardiovascular prevention goal. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2779-85. doi: 10.1016/j.jacc.2014.04.009. Epub 2014 May 7. PMID 24814489